CLINICAL TRIAL: NCT01604733
Title: Centralized Pan-Middle East Survey on the Undertreatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-EG-CRE-2010/01
Record Dates: First submitted 2012-05-21; First posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Multi-Center Survey; patients currently on lipid-lowering pharmacological treatment; level of Control of Hypercholesterolemia in Egypt
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HYPERCHOLESTEROLEMIC PATIENTS

SUMMARY:
Study objective is to evaluate the level of control of hypercholesterolemia in Egypt in patients taking lipid lowering agents for at least 3 months ( with no drug change or dose amendment for a minimum of 6 weeks).

DETAILED DESCRIPTION:
Centralized Pan-Middle East Survey on the Undertreatment of Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above on current lipid lowering drug for at least 3 months with no dose change for a minimum of 6 weeks
* Subject must provide informed consent and comply with the survey procedures

Exclusion Criteria:

* Less than 18 years less than 3 months on antidyslipidemic agent Subjects who are unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients on lipid-lowering treatment reaching the LDL-C goals according to the NCEP ATP III/ updated 2004 NCEP ATP III , overall and by country | 24 weeks

SECONDARY OUTCOMES:
The proportion of patients on lipid-lowering treatment reaching the LDL-C goals according to the NCEP ATP III/ updated 2004 NCEP ATP III , in the following sub-populations: - primary/secondary prevention patients and with metabolic syndromes | 24 weeks
The proportion of patients on lipid-lowering treatment reaching the LDL-C goals according to the Third Joint European Task Force guideline, in the following sub-populations: - primary/secondary prevention patients and with metabolic syndromes | 24 weeks
Determinants (e.g. patient and physician characteristics , country-specific guidelines or recommendations) for undertreatment of hypercholesterolemia | 24 weeks
Physician characteristics associated with the allocation of treatment regimen. | 24 weeks
The proportion of patients on lipid-lowering treatment reaching the non HDL-C goals according to the NCEP ATP III/ updated 2004 NCEP ATP III , in the sub-population patients with fasting triglycerides<200 mg/d | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohie E Sherif, MD, Study Chair — Ethical committee, Faculty of medicine, Alexandria University